CLINICAL TRIAL: NCT05541172
Title: Testosterone Undecanoate Replacement Therapy in Boys With Pubertal Delay or Confirmed Hypogonadism
Status: Recruiting | Type: Observational
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Collaborators: National Agency for Scientific and Technological Promotion, Argentina (Other)
Responsible Party: Principal Investigator, Dr Rodolfo Rey, Director of CEDIE, Hospital de Niños R. Gutierrez de Buenos Aires
Other Study IDs: CEI 21-07
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Delayed Puberty; Male Hypogonadism
MeSH Terms: conditions — Puberty, Delayed; Eunuchism | interventions — testosterone undecanoate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Testosterone Undecanoate — Testosterone undecanoate (1000 mg/4 ml) will be administered at a dose of 1 ml every 12 weeks for 6 months, 2 ml every 12 weeks for 6 months, 3 ml every 12 weeks for 6 months and 4 ml every 12 weeks for 6 months.

SUMMARY:
The absence of clinical signs of pubertal maturation, i.e. pubertal delay, is a relatively frequent reason for consultation in boys. In cases where it is necessary, the treatment to be established is the administration of testosterone with the aim of provoking the development of secondary sexual characteristics and optimizing growth.

Currently, the most commonly used treatment is empirical, with im testosterone enanthate at increasing doses (from 50 mg every 4 weeks up to 250 mg every 4 weeks) over a period of 2 to 3 years. The pharmacokinetic profile has not been described to see if it mimics the physiological progressive increase in testosterone levels occurring during normal puberty. In adults, testosterone enanthate shows supraphysiological serum testosterone the first week after, with a progressive drop to subphysiological levels in the fourth week.

Testosterone undecanoate is used in adults at a dose of 1000 mg im every 12 weeks, as equivalent to testosterone enanthate 250 mg every 4 weeks.Serum levels of testosterone show a profile within physiological ranges. Testosterone undecanoate im has not been tested in adolescents.

Hypothesis: The hypothesis of this work is that the initial administration of 1 ml (~250 mg) of testosterone undecanoate (1000 mg/4 ml) via im every 12 weeks for 6 months, with a progressive increase of 1 ml (~250 mg) every 6 months until reaching 4 ml (1000 mg) per dose is safe and effective in causing normal progression of secondary sex characteristics and growth spurt in boys with pubertal delay.

The primary specific objectives are to determine, in boys with pubertal delay: (a) if a treatment regimen of testosterone undecanoate (1000 mg/4 ml), with an initial dose of 250 mg every 12 weeks and subsequent increase up to 1000 mg every 12 weeks over 2 years (increasing 250 mg every 6 months) induces a progression in the development of secondary sexual characteristics and growth spurt commensurate with those of normal pubertal development, and (b) the safety of the administration of increasing doses of im testosterone undecanoate.

DETAILED DESCRIPTION:
Introduction: The absence of clinical signs of pubertal maturation, i.e. pubertal delay, is a relatively frequent reason for consultation in boys. In cases where it is necessary, the treatment to be established is the administration of testosterone with the aim of provoking the development of secondary sexual characteristics and optimizing growth.

Problem: Currently, the most commonly used treatment is empirical, with im depot testosterone at increasing doses over a period of 2 to 3 years. The most commonly used formulation, testosterone enanthate, comes in ampoules of 250 mg in 1 ml of vehicle. The usual administration regimen begins with approximately 50-60 mg im every 4 weeks (1/4 of the ampoule), increasing the dose by approximately 50-60 mg (1/4 ampoule) every 6 months until the full dose of 250 mg (1 ampoule) is reached every 4 weeks. The pharmacokinetic profile has not been described to see if it mimics the physiological progressive increase in testosterone levels at normal puberty. The pharmacokinetic profile of testosterone enanthate in adults shows supraphysiological serum testosterone concentrations the first week after the medication is administered, with a progressive drop to subphysiological levels in the fourth week.

In adults, testosterone undecanoate is used as a first-line medication. Its presentation in ampoules with 1000 mg in 4 ml, of im administration every 12 weeks, is considered equivalent to testosterone enanthate 250 mg every 4 weeks. In adults, the circulating levels of testosterone obtained with the formulation of testosterone undecanoate show a profile within physiological ranges, more stable between doses than that observed with testosterone enanthate. Testosterone undecanoate im has not been tested in adolescents.

Hypothesis: The hypothesis of this work is that the initial administration of 1 ml (~250 mg) of testosterone undecanoate (1000 mg/4 ml) via im every 12 weeks for 6 months, with a progressive increase of 1 ml (~250 mg) every 6 months until reaching 4 ml (1000 mg) per dose is safe and effective in causing normal progress in pubertal development of secondary sex characteristics and growth in males with pubertal delay.

Objective: The general objective of this study is to evaluate whether a quarterly administration regimen of im testosterone undecanoate, in boys with anorchia, hypogonadism or pubertal delay induces the progression in the development of secondary sexual characteristics, the speed of growth and the acquisition of bone mass in accordance with physiological pubertal development, and maintain blood testosterone levels similar to those seen during spontaneous pubertal maturation.

The primary specific objectives are to determine, in boys with pubertal delay:

1. If a treatment regimen of testosterone undecanoate (1000 mg/4 ml) im, with an initial dose of 1 ml (~250 mg) every 12 weeks (stage 1: weeks 1-24), 2 ml (~500 mg) every 12 weeks (stage 2: weeks 25-48), 3 ml (~750 mg) every 12 weeks (stage 3: weeks 49-72) and 4 ml (100 0 mg) every 12 weeks (stage 4: weeks 73-96), is accompanied by progress in the development of secondary sexual characteristics and growth rate commensurate with those of normal pubertal development.
2. The safety of the administration of increasing doses of im testosterone undecanoate, through the evaluation of biochemical parameters (see below) and bone age progress.

The secondary specific objectives are:

1. To assess whether blood testosterone levels are maintained at levels within established physiological limits, for 12 weeks after administering the dose of testosterone undecanoate im.
2. To explore the changes occurring in the pituitary-gonadal axis and bone mass of boys with pubertal delay who are treated with increasing doses of im testosterone undecanoate.

Design and methods: An intervention study will be carried out, with prospective longitudinal follow-up of a cohort of boys with anorchia, hypogonadism or pubertal delay.

Testosterone undecanoate (1000 mg/4 ml) will be administered at a dose of 1 ml every 12 weeks for 6 months, 2 ml every 12 weeks for 6 months, 3 ml every 12 weeks for 6 months and 4 ml every 12 weeks for 6 months.

Progression commensurate with normal pubertal development shall be considered to exist if the clinical evaluation detects a Tanner stage G2 or G3 and PH2 or PH3 at the end of the first 6 months, G3 or G4 and PH3 or PH4 at the end of the first year, G3 to G5 and PH3 to PH5 after 18 months, and G4 or G5 and PH4 to PH6 at the end of 2 years. The proportion of patients with the hypothesized progression will be calculated. The therapeutic scheme shall be considered satisfactory if this proportion is ≥80%.

For growth, progression in line with normal pubertal maturation shall be considered if the clinical evaluation detects a height velocity of 6 to 10 cm/year at the end of the first year and 8 to 14 cm/year at the end of the second year. The proportion of patients with the hypothesized progression will be calculated. The therapeutic scheme shall be considered satisfactory if this proportion is ≥80%.

The number and type of adverse events at each visit will be reported. Changes in hormone levels of the pituitary-gonadal axis and bone mass will be analyzed.

Sample size: For this study, estimating that 80% of patients will have a development of secondary sexual characteristics within the range expected for each stage after the administration of 1, 2, 3 or 4 ml of testosterone undecanoate im every 12 weeks, it will be necessary to analyze 27 individuals to provide a conclusion with an accuracy of 15%. Accepting a maximum loss of 20% during follow-up, 34 patients should be recruited into the study.

Statistical analysis: A descriptive statistical report of the quantitative variables will be carried out, using mean and standard deviation or median and interquartile range according to whether they follow a normal distribution, evaluated by the Shapiro-Wilk test. The proportions will be reported by further calculating the 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Males between 13 and 18 years old without signs of pubertal development, or between 12 and 18 years old with a confirmed diagnosis of anorchia or hypogonadism.
* Normal male configuration of the external genitalia for Tanner G1 stage, with or without palpable testicles, as defined in 4.5.
* As appropriate, assent/consent of the patient and their parents or guardians.

Exclusion Criteria:

* Bone age < 11 years.
* Allergy to the medication of the study.

Ages: 12 Years to 18 Years | Sex: Male
Age Groups: Child, Adult
Study Population: The target population includes boys diagnosed with anorchia, hypogonadism, or CDGP requiring testosterone treatment.
  All eligible patients who present consecutively until the sample size is completed will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression in the development of secondary sexual characteristics | 2 years
  Progression of pubertal stages will be considered as in line with normal maturation if the clinical evaluation detects Tanner G2 or G3 and pubic hair (PH)2 or PH3 at the end of stage 1 (visit 8), G3 or G4 and PH3 or PH4 at the end of stage 2 (visit 14), G3 to G5 and PH3 to PH5 at the end of stage 3 (visit 20 ), and G4 or G5 and PH4 to PH6 at the end of stage 4 (visit 26).
  The proportion of patients with progression as hypothesized will be calculated. The therapeutic regimen shall be considered satisfactory if this proportion is ≥80%
Progression in the speed of growth | 2 years
  Height velocity calculated as Δ stature (cm)/Δ time (months). Progression will be considered as in line with normal growth if the clinical evaluation detects a height velocity of 6 to 10 cm/year at the end of stage 2 (visit 14) and 8 to 14 cm/year at the end of stage 4 (visit 26). The proportion of patients with progression as hypothesized will be calculated. The therapeutic regimen shall be considered satisfactory if this proportion is ≥80%.

SECONDARY OUTCOMES:
Testosterone concentration in serum | 2 years
  Values will be considered to be within the target range if they are between 20 and 80 ng/dl in visits 4 and 7, between 100 and 180 ng/dl in visits 10 and 13, between 200 and 300 ng/dl in visits 16 and 19 and between 350 and 900 ng/dl in visits 22 and 25.

OTHER OUTCOMES:
Adverse events | 2 years
  The number and type of adverse events at each visit. The ratio Δ bone age (months)/Δ chronological age (months). Bone age will be considered to be accelerated if an increase of more than 12 months is found for every 6-month period of treatment, between visit 1 and visit 8, between visit 8 and visit 14, or between visit 14 and visit 20.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Rey, Study Director — Hospital de Niños R. Gutierrez
Locations (1):
- Rodolfo Rey, Buenos Aires, Distrito Federal, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT05541172/Prot_SAP_000.pdf